CLINICAL TRIAL: NCT02415426
Title: Metacognitive Training Program With Depression
Acronym: DMKT
Status: Terminated | Type: Observational
Sponsor: Psychiatric University Hospital, Zurich (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Egemen Savaskan, Prof. Dr. med., Psychiatric University Hospital, Zurich
Other Study IDs: D-MKT - 2014-0421
Record Dates: First submitted 2015-03-26; First posted 2015-04-14 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

INTERVENTIONS:
Behavioral: Metacognitive Training Program during mild to moderate depression — Diagnostic and therapeutical interventions are not part of this study. As part of this study, the change of cognitive and psychosocial achievement/behavior in patients with mild to moderate depression after taking part in the training program is being investigated. The training program seeks to enable group members to recognize and correct the often automatic and unconscious thought patterns that accompany depression, in part by viewing this depressive thought process at a distance (i.e., depersonalizing). In addition, dysfunctional assumptions about one's thought processes, as well as dysfunctional coping-strategies (i.e., thought suppression, rumination as problem-solving) are targeted (Lena Jelinek & Steffen Moritz, http://clinical-neuropsychology.de/metacognitive_training_for_depression.html).

SUMMARY:
The participants of this study have been diagnosed with mild to moderate depression with no evidence of suicidal actions prior to recruitment. All recruited subjects receive standard therapy and participate in a metacognitive training program (D-MKT) independently of study participation. Diagnostic and therapeutical interventions are not part of this study. As part of this study, the change of cognitive and psychosocial achievement/behavior in patients with mild to moderate depression after taking part in the training program is being investigated. The training program seeks to enable group members to recognize and correct the often automatic and unconscious thought patterns that accompany depression, in part by viewing this depressive thought process at a distance (i.e., depersonalizing). In addition, dysfunctional assumptions about one's thought processes, as well as dysfunctional coping-strategies (i.e., thought suppression, rumination as problem-solving) are targeted (Lena Jelinek & Steffen Moritz, http://clinical-neuropsychology.de/metacognitive_training_for_depression.html). Within this study the cognitive and psychosocial behaviour changes are being investigated by neuropsychological assessment as well as questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the Metacognitive Training Program
* Subjects with an age over 55 years and a diagnosed mild to moderate depression without psychotic Symptoms (F32, F33)
* Subjects have to be able to understand verbal and written information regarding treatment and procedures of the study.
* Subjects have to be able to understand and perform verbal and written tasks (cognitive tests/questionnaires).
* No evidence of suicidal tendency

Exclusion Criteria:

* Taking of medication or drugs that could influence cognition
* Diseases that prevent the subject from giving consent to this study or affect the collaboration during the examination
* Major and/or unstable physical diseases
* Strongly impaired vision/eye diseases
* Psychotic or manic symptoms
* Benzodiazepine addiction/dependency
* Suicidal tendency

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients from our ambulatorium
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2015-06; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Improvement of depression as measured by Becks Depression Inventory (BDI) | 14 months
Improvement of depression as measured by Hamilton Depression Scale (HAMD) | 14 months
Improvement of self-esteem as measured by Rosenberg Self-esteem Scale (RSE) | 14 months
Improvement of dysfunctional coping strategies as measured by 10-Item-Version of the Response Styles Questionnaire in German (RSQ-D) | 14 months
Improvement of dysfunctional coping strategies as measured by Dysfunctional Attitude Scale (DAS) | 14 months
Improvement of satisfaction and subjective well-being as measured by World Health Organization Quality of Life - short version (WHOQOL-BREF) | 14 months
Improvement of metacognitive thinking as measured by Metacognitions Questionnaire (MCQ) | 14 months
Improvement of cognition as measured by Consortium to Establish a Registry for Alzheimer's Disease (CERAD-Plus) | 14 months
Improvement of cognition as measured by 5-Point Test | 14 months
Improvement of cognition as measured by Regensburger Wortflüssigkeitstest (RWT) | 14 months
Improvement of cognition as measured by Tower of London | 14 months
Improvement of cognition as measured by Wechsler Memory Scale Revised (WMS-R) | 14 months
Improvement of cognition as measured by Trail Making Test (TMT) | 14 months
Improvement of cognition as measured by Wechsler Adult Intelligence Scale (WAIS-IV) | 14 months
Improvement of cognition as measured by Verbaler Lern- und Merkfähigkeitstest (VLMT) | 14 months
Improvement of cognition as measured by Testbatterie zur Aufmerksamkeitsprüfung (TAP) | 14 months
Improvement of cognition as measured by MWT | 14 months
Improvement of cognition as measured by Cartoon Test | 14 months
Improvement of cognition as measured by Faux Pas Test | 14 months

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik für Alterspsychiatrie, Gerontopsychiatrisches Zentrum Hegibach, Zurich, Switzerland